CLINICAL TRIAL: NCT03152695
Title: To Evaluate the Safety and Efficacy of High-intensity Focused Ultrasound (HIFU) for the Symptom Relief of Inoperable Abdominal Tumors
Brief Title: High-intensity Focused Ultrasound (HIFU) for the Symptom Relief of Inoperable Abdominal Tumors
Acronym: HIFU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201701032DIPD
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-01

CONDITIONS: Symptomatic Abdominal Tumour

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-intensity focused ultrasound therapy (Experimental): Abdominal MRI will be used to target the tumor, and the tumor will be divided into slices with 5mm separation using MR images. By scanning the HIFU beam in successive sweeps from the deep to the shallow regions of the tumor.
  Interventions: Device: High-intensity focused ultrasound

INTERVENTIONS:
Device: High-intensity focused ultrasound — Local tumor ablation by ArcBlate (EpiSonica, Taiwan) will be performed, and the entire procedure will be monitored by MRI

SUMMARY:
High-intensity focused ultrasound (HIFU), a recently developed tumor ablation equipment, can be a non-invasive treatment for solid tumors. The principle of HIFU is physically focus the ultrasound point on the biological tissue to form high-intensity ultrasound focus, and kill tumor cells by the thermal effects, mechanical effects and acupuncture effects of the high-intensity ultrasound.

DETAILED DESCRIPTION:
The clinical recommendations for unresectable malignant tumors, which cause pain and other symptoms, are chemotherapy or local radiation therapy to delay tumor progression, improve life quality and prolong survival, while there is no other effective recommendations for benign tumors., Local ablation, such as radiofrequency ablation (RFA), is expected to be another therapeutic option for tumors that cannot be surgically resected. However, the main drawback of radiofrequency ablation is that its puncture invasion can sometimes cause bleeding or tumor metastasis. The peripheral blood vessels can also cause poor ablation, therefore; RFA is limited to small liver cancer treatment.

High-intensity focused ultrasound (HIFU), a recently developed tumor ablation equipment, can be a non-invasive treatment for solid tumors. The principle of HIFU is physically focus the ultrasound point on the biological tissue to form high-intensity ultrasound focus, and kill tumor cells by the thermal effects, mechanical effects and acupuncture effects of the high-intensity ultrasound.

Under the real-time magnetic resonance imaging system and a variety of appropriate scanning to move the focused ultrasound in the treatment area to kill the tumor. The tumor that is killed will gradually absorb and fibrosis in the body. There is no significant invasion due to it is without penetrating the needle into body. This system has been approved and certificated for the use of soft tissue ablation by Taiwan Food and Drug Administration (TFDA) in 2016. The main participants of this study are patients who have benign and malignant tumors in the abdominal cavity with tumor-related symptoms and not suitable for surgical resection. The investigators will conduct HIFU, observe whether there is any complications after surgery. Moreover, the investigators will notice the tumor response after a month and track the survival rate to verify the feasibility and advantages of HIFU for clinical use.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must meet all of the following inclusion criteria to be eligible for this study:

1. Eligible patients with symptomatic intra-abdominal tumor including liver, pancreas, bile duct and retroperitoneal tumors will be enrolled for study.
2. The criteria for unresectability included evidence of distant metastatic disease, involvement of the major vessels and high risk of functional insufficiency after tumor excision.
3. Eastern Cooperative Oncology Group (ECOG) score of 0-1,
4. American Society of Anaesthesiologists (ASA) score ≤ 3,
5. Adequate bone marrow, liver and renal function (1). Platelet count ≥ 100 K/Μl(2). Total bilirubin ≦ 5 mg/dL(3). Alanine transaminase (ALT) and aspartate transaminase (AST) < 5 x upper limit of normal (4). Prothrombin time (PT)- international normalized ratio (INR) ≦ 2.0 (5). Serum creatinine ≦ 2 x upper limit of normal
6. Prior Informed Consent Form
7. Life expectancy of at least 3 months.

Exclusion Criteria:

* Patients presenting with any of the following will not be enrolled into this study:

  1. The tumor cannot be visualized by abdominal MRI.
  2. No suitable approach route for ultrasound toward tumor under image evaluation, for example scar formation, bowel gas, bone within the ultrasound window.
  3. Women who are pregnant.
  4. The patients had received treatment with an investigational agent/ procedure within 30 days prior to this study.
  5. Arterial calcification was noted within the treatment window of ultrasound.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of tumour response | 1 month after treatment
  Evaluation of tumour response according to the modified RECIST criteria by sequencing CT or MR imaging

SECONDARY OUTCOMES:
To evaluate the overall survival | within one year
  using Common Terminology Criteria for Adverse Events (CTCAE). Version 4.0 and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Wen Huang, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan